CLINICAL TRIAL: NCT03845023
Title: Phase 2, Placebo-Controlled, Parallel Group Dose-Finding Study to Evaluate the Efficacy and Safety of Three Dose Levels of AD036 in Adults With Obstructive Sleep Apnea
Brief Title: Trial of AD036 in Obstructive Sleep Apnea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Apnimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APN-002
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Results first posted 2023-01-17 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — (Lys-Gly)(5)cyclo(75-82)MBP(74-85)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 2-Night at Home (Placebo Comparator): An initial 2-night, at-home blinded baseline period in which all subjects received placebo
  Interventions: Drug: Placebo
- 3-Night Run In (Experimental): AD036 Dose 1 (Low Dose: 25/5) or Placebo
  Interventions: Drug: AD036 Dose 1; Drug: Placebo
- 7-Night (Experimental): A 7-night treatment period in which subjects received the treatment to which they were randomized, i.e., 1 of the 3 different fixed-dose combinations of drugs, or placebo
  Interventions: Drug: AD036 Dose 1; Drug: AD036 Dose 2; Drug: AD036 Dose 3; Drug: Placebo
- End of Study (No Intervention): End of Study Visit

INTERVENTIONS:
Drug: AD036 Dose 1 — AD036 Dose 1 oral capsule administered before sleep
  Other Names: 25/5
  Arms: 3-Night Run In; 7-Night
Drug: AD036 Dose 2 — AD036 Dose 2 oral capsule administered before sleep
  Other Names: 75/1.5
  Arms: 7-Night
Drug: AD036 Dose 3 — AD036 Dose 3 oral capsule administered before sleep
  Other Names: 75/5
  Arms: 7-Night
Drug: Placebo — Placebo oral capsule administered before sleep
  Arms: 2-Night at Home; 3-Night Run In; 7-Night

SUMMARY:
This is a randomized, double blind, placebo-controlled, repeat-dose, parallel arm, outpatient and inpatient phase 2 clinical study to examine the efficacy and safety of three dose levels of AD036 versus placebo in patients with obstructive sleep apnea.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled, repeat-dose, parallel arm, outpatient and inpatient, multicenter, dose-finding study of the combination of atomoxetine and oxybutynin in adults with OSA documented by polysomnography (PSG).

Approximately 140 subjects were to be randomized 1:1:1:1 to receive 1 of 3 different fixed-dose combinations of oxybutynin and atomoxetine or matching placebo.

For all subjects, the study consisted of:

* A screening and baseline period in which subjects' eligibility was determined
* An initial 2-night, at-home blinded baseline period in which all subjects received placebo
* A 3-night, run-in period in which subjects received:

  * Low-dose combination for subjects randomized to one of the 3 study treatment arms
  * Placebo for subjects randomized to the placebo treatment arm
* A 7-night treatment period in which subjects received the treatment to which they were randomized, i.e., 1 of the 3 different fixed-dose combinations of drugs, or placebo
* An end of study visit

ELIGIBILITY:
Male participants between 25 to 65 years of age or female participants between 25 to 70 years of age.

Key Inclusion Criteria:

* AHI ≥ 20 based on screening polysomnography
* Epworth Sleepiness Scale (ESS) score ≥ 4 for participants not using CPAP
* Previous surgical treatment for OSA is allowed if ≥ 1 year prior to enrollment

Key Exclusion Criteria:

* Clinically significant craniofacial malformation.
* Clinically significant cardiac disease (e.g., rhythm disturbances, coronary artery disease or cardiac failure) or hypertension requiring more than 2 medications for control.
* Clinically significant neurological disorder, including epilepsy/convulsions.
* Positive screen for drugs of abuse or substance use disorder as defined in DSM-V within 24 months prior to Screening Visit.
* A significant illness or infection requiring medical treatment in the past 30 days.
* Women who are pregnant or nursing.
* History of using oral or nasal devices for the treatment of OSA may enroll as long as the devices are not used during participation in the study.
* History of using devices to affect participant sleeping position for the treatment of OSA, e.g. to discourage supine sleeping position, may enroll as long as the devices are not used during participation in the study.
* Treatment with strong cytochrome P450 3A4 (CYP3A4) inhibitors, strong cytochrome P450 2D6 (CYP2D6) inhibitors, or monoamine oxidase inhibitors (MAOI) within 14 days of the start of treatment, or concomitant with treatment.
* Use of another investigational agent within 90 days or 5 half-lives, whichever is longer, prior to dosing.
* ESS total score > 18.
* Central apnea index > 5/hour on baseline PSG.
* Periodic limb movement arousal index >15/hour on baseline PSG.
* Hepatic transaminases >3X the upper limit of normal (ULN), total bilirubin >2X ULN (unless confirmed Gilbert syndrome), serum creatinine >2X ULN.
* <6 hours typical sleep duration.
* Night- or shift-work sleep schedule.
* Employment as a commercial driver or operator of heavy or hazardous equipment.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Farkas, MD, Study Director — Apnimed
Locations (12):
- United States (12):
  - Pulmonary Associates, Glendale, Arizona
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Stanford Sleep Medicine, Redwood City, California
  - SDS Clinical Trials, Inc., Santa Ana, California
  - Santa Monica Clinical Trials, Santa Monica, California
  - Northwestern University, Chicago, Illinois
  - Norton Clinical Research Group, Louisville, Kentucky
  - The Center for Sleep and Wake Disorders, Chevy Chase, Maryland
  - Sleep Medicine & Research Center, St. Luke's Hospital, Chesterfield, Missouri
  - Clinilabs Drug Development Corporation, New York, New York
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Sleep Therapy & Research Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 12 clinical sites (hospitals and sleep centers). The study population consisted of male and female subjects between 25 and 65 years of age, inclusive, with OSA documented by PSG. Overall study duration was up to 8 weeks. Dosing of the study treatment was to occur approximately 30 minutes prior to bedtime. Subjects who withdrew from the study were not replaced.
Groups:
- Placebo: Placebo oral capsule administered orally at bedtime
- AD036 Dose 1: AD036 Dose 1 (Low Dose 25/5) administered orally before bedtime
- AD036 Dose 2: 75/1.5 administered orally at bedtime.
- AD036 Dose 3: AD036 75/5 administered orally at bedtime
Period: Placebo Run-In Period (2 Nights)
Arm/Group | Placebo | AD036 Dose 1 | AD036 Dose 2 | AD036 Dose 3
Started | 36 | 36 | 34 | 34
Completed | 36 | 36 | 34 | 34
Not Completed | 0 | 0 | 0 | 0
Period: Low Dose Run-In (3 Nights)
Arm/Group | Placebo | AD036 Dose 1 | AD036 Dose 2 | AD036 Dose 3
Started | 36 | 36 | 34 | 34
Completed | 36 | 36 | 34 | 34
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period (7 Nights)
Arm/Group | Placebo | AD036 Dose 1 | AD036 Dose 2 | AD036 Dose 3
Started | 36 | 36 | 34 | 34
Completed | 36 | 36 | 34 | 34
Not Completed | 0 | 0 | 0 | 0
Period: Follow-Up (14 Days)
Arm/Group | Placebo | AD036 Dose 1 | AD036 Dose 2 | AD036 Dose 3
Started | 36 | 36 | 34 | 34
Completed | 35 | 36 | 33 | 33
Not Completed | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Data presented is from the safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AD036 Dose 1 | AD036 Dose 2 | AD036 Dose 3 | Total
Number analyzed (Participants) | 36 | 36 | 34 | 34 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 35 | 33 | 31 | 132
  >=65 years | 3 | 1 | 1 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 7 | 12 | 42
  Male | 25 | 24 | 27 | 22 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 3 | 4 | 11
  Not Hispanic or Latino | 34 | 34 | 31 | 30 | 129
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 3 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 15 | 10 | 8 | 11 | 44
  White | 18 | 25 | 23 | 21 | 87
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
BMI (kg/m^2) [Median (Full Range); unit: kg/m^2] | 32.930 [22.74 to 40.30] | 33.445 [22.30 to 39.36] | 32.555 [20.64 to 40.17] | 33.170 [22.19 to 39.82] | 32.745 [20.64 to 40.30]

OUTCOME MEASURES:

1. Primary Outcome: Apnea Hypopnea Index (AHI)
Description: Number of participants with ≥50% reduction in apnea hypopnea index (AHI). AHI is the average number of apneas and hypopneas a person experiences each hour during sleep, to register as an event an apnea or hypopnea must last at least 10 seconds or longer. To measure this, doctors divide the total number of apneic and hypopneic events by the total number of hours the person was asleep.
Time Frame: 10 days
Population: All randomized subjects were included in the mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AD036 Dose 1 | AD036 Dose 2 | AD036 Dose 3
Number analyzed (Participants) | 36 | 36 | 34 | 34
Participants
  Yes (subjects that had a 50% reduction in AHI) | 3 | 2 | 6 | 8
  No (subjects that did not have a 50% reduction in AHI) | 33 | 34 | 28 | 26

ADVERSE EVENTS:
Time Frame: Adverse events were collected over an 8 month period
Description: The study analysis did not analyze data by period. AEs were reported for the safety analysis by number and percent for treatment group only.
Arm/Group | Placebo | AD036 Dose 1 | AD036 Dose 2 | AD036 Dose 3
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/104 | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/140 | 1/104 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 7/140 | 13/104 | 16/34 | 14/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=140) | AD036 Dose 1 (N=104) | AD036 Dose 2 (N=34) | AD036 Dose 3 (N=34)
Acute Kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not Related
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=140) | AD036 Dose 1 (N=104) | AD036 Dose 2 (N=34) | AD036 Dose 3 (N=34)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 6 (6) | 2 (2) | 8 (8)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 5 (5)
dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
headache (Nervous system disorders) | 3 (3) | 4 (4) | 7 (7) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Poor Quality Sleep (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 5 (5) | 3 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Middle Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Urinary Hesitation (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Urine output decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs agreed that because the Study is part of a Multi-center Study, individual publication could not be made until the publication of the Multi-center study results, notification that that a Multi-center publication was not planned, or after 18 months had passed.

DOCUMENTS (2):
  • Study Protocol (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/23/NCT03845023/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT03845023/SAP_001.pdf